CLINICAL TRIAL: NCT05899725
Title: The Efficacy and Safety of Corticosteroids in Combination With Biological Agents in the Management of Severe Immune Related Adverse Events Cohort A: The Efficacy and Safety of Corticosteroids or Corticosteroids Combination With Ruxolitinib in Patients With Severe Checkpoint Inhibitor Pneumonia
Brief Title: The Efficacy and Safety of Corticosteroids in Combination With Ruxolitinib in the Management of Checkpoint Inhibitor Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wang mengzhao, Chief Director of Department of Respiratory and Critical Care Medicine, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K22C2678
Record Dates: First submitted 2023-06-03; First posted 2023-06-12 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Severe Checkpoint Inhibitor Pneumonitis
MeSH Terms: interventions — Adrenal Cortex Hormones; ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: severe CIP with the treatment of corticosteroids (Active Comparator): severe CIP with the treatment of corticosteroids
  Interventions: Drug: Corticosteroids
- Cohort 2: severe CIP with the treatment of corticosteroids and Ruxolitinib (Experimental): severe CIP with the treatment of corticosteroids and Ruxolitinib
  Interventions: Drug: Corticosteroids and Ruxolitinib

INTERVENTIONS:
Drug: Corticosteroids — Initial dosage of corticosteroids is no less than predinisone 1mg/kg/d or other corticosteroids with equal equivalence
  Arms: Cohort 1: severe CIP with the treatment of corticosteroids
Drug: Corticosteroids and Ruxolitinib — Initial dosage of corticosteroids is no less than predinisone 1mg/kg/d or other corticosteroids with equal equivalence, add-on oral Ruxolitinib 5mg twice a day for 2 weeks, following with Ruxolitinib
  Arms: Cohort 2: severe CIP with the treatment of corticosteroids and Ruxolitinib

SUMMARY:
This study is a prospective multicenter randomized controlled Interventional study, to assess the clinical efficacy and safety of corticosteroids compared to corticosteroids in combination with Ruxolitinib in the treatment of severe checkpoint inhibitor pneumonitis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old≤ Aged ≤80 years old.
2. Diagnosis of malignancy.
3. Malignant tumors initially treated with immune checkpoint inhibitors (antibodies targeting PD-1, PD-L1, CTLA-4, or new immune checkpoint inhibitors) in combination with or without chemotherapy.
4. Diagnosis of grade 3 or 4 CIP: CIP severity at CTCAE grade 3 or 4.
5. Patients who and whose family members understand the study protocol, are willing to participate in the study and could provide written informed consent.

Exclusion Criteria:

1. Predicted life expectancy<12 weeks.
2. Any evidence of active or uncontrolled viral infection, including hepatitis B, hepatitis C and human immunodeficiency virus (HIV), or any clinical signs of bacterial, other viral, parasitic or fungal infection requiring treatment.
3. malignancy progression.
4. Patients with other serious complications that may affect safety or adherence judged by the investigator.
5. Any significant clinical and laboratory abnormalities judged by investigator that affect the safety evaluation.
6. Patients can't fully understand the study protocol, arrangement and other study-related elements.
7. Patients with evidence of severe liver or kidney dysfunction judged by investigator unsuitable for enrolment.
8. Women who are pregnant, breast feeding or unable to use effective contraception during the study period and for 3 months after the completion.
9. Patients who cannot comply with study treatment and follow-up according to the trial protocol.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with dosage of corticosteroids no more than 10mg daily at improvement to CIP with CTCAE grade 1. | 8 weeks
  Proportion of patients with dosage of corticosteroids no more than 10mg daily at improvement to CIP with CTCAE grade 1.

SECONDARY OUTCOMES:
Mortality | 8 weeks
  Mortality of severe CIP patients at 8 weeks.
Proportion of invasive ventilator assisted respiration | 8 weeks
  Proportion of invasive ventilator assisted respiration treatment for severe CIP patients at 8 weeks.
Incidence of pulmonary infection | 8 weeks
  Incidence of pulmonary infection in severe CIP patients in 8 weeks.
Total corticosteroids usage | 8 weeks.
  Total corticosteroids usage for severe CIP patients in 8 weeks.
The incidence of treatment with immunosuppressants and the incidence of treatment with IVIG | 8 weeks.
  The incidence of treatment with immunosuppressants and the incidence of treatment with IVIG for severe CIP patients in 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory Medicine, Peking Union Medical College Hospita, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided